CLINICAL TRIAL: NCT06440590
Title: Supra-Pectineal Quadrilateral Buttress Plating Versus Infra-pectineal Plating in Management of Quadrilateral Plate Fractures: A Randomized Controlled Trial
Brief Title: Supra-Pectineal QLS Plating Vs Infra-pectineal Plating in Management of Quadrilateral Plate Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Islam Moussa, lecturer of orthopedic surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU R66/2023
Record Dates: First submitted 2024-05-26; First posted 2024-06-04 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Evaluation of QL Buttress Plating in QLP Fracture Fixation
Keywords: quadrilateral plate fractures; anterior column fractures; associated both column fractures; infra-pectineal plating; supra-pectineal quadrilateral buttress plating

STUDY DESIGN:
Intervention Model Description: An independent doctor created the randomization sequence using Excel 2016 (computerized random numbers) with a 1:1 allocation via random block sizes of 2, 4, and 6; he assigned the sample numbers equally to each group and assigned the block. Patients and physicians allocated to each intervention group were aware of the allocation; however, the data analysts and the outcome assessors were kept blinded to the allocation. The investigators prospectively carried out this study on 30 patients with quadrilateral plate fractures between February 2022 and June 2023 that met our inclusion criteria. The independent doctor allocated the 30 cases to two groups: Group A (15 cases): supra-pectineal quadrilateral buttress plating, group B (15 cases): Infra-pectineal plating
Who Masked: Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor) Patients and physicians allocated to each intervention group were aware of the allocation; however, the data analysts and the outcome assessors were kept blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supra-pectineal quadrilateral buttress plating (Active Comparator): Patients treated by supra-pectineal quadrilateral buttress plating through anterior intrapelvic approach
  Interventions: Procedure: suprapectineal quadrilateral buttress plating
- Infrapectineal plating (Active Comparator): Patients treated by infra-pectineal conventional plating applied on the medial wall through anterior intrapelvic approach
  Interventions: Procedure: Infra-pectineal plating

INTERVENTIONS:
Procedure: suprapectineal quadrilateral buttress plating — 15 cases will undergo anatomical supra-pectineal quadrilateral plate
  Arms: supra-pectineal quadrilateral buttress plating
Procedure: Infra-pectineal plating — 15 cases will undergo conventional manually contoured infra-pectineal plate
  Arms: Infrapectineal plating

SUMMARY:
The investigators conducted such a prospective randomized controlled study aiming to reach a satisfactory outcome and to compare supra-pectineal QL buttress plating versus infra-pectineal for management of anterior column with or without posterior hemi-transverse component and quadrilateral plate involvement.

DETAILED DESCRIPTION:
Our hypothesis was that supra-pectineal quadrilateral buttress plating provides much more rigid fixation and a strong buttress for medial wall migration, also it could correlate with a better functional and radiological outcome. However, there is a lack of knowledge in the prospective assessment of functional and radiological outcomes and follow up of postoperative complications of supra-pectineal quadrilateral buttress plating versus infra-pectineal plating in fixation of QLS and to our knowledge, it will be the first study to include such measures of outcome together in a prospective randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

* Anterior column fracture acetabulum with QLS involvement
* Anterior column posterior hemi-transverse fracture acetabulum with QLS involvement
* Age between 16-60 years' old

Exclusion Criteria:

* Open fractures
* Associated pelvic ring injuries that require intervention
* Associated internal organ injuries that require intervention
* Age less than 14 years and older than 60 years

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Excellent, very good, Good, Average or Poor functional outcomes using Modified Merle d'Aubigné scoring system | one-year post-operative
  Clinical assessment was done via Modified Merle d'Aubigné scoring system that was calculated at each follow-up visit (out of 18) and presented the mean value; the score evaluates three factors: pain, mobility & ability to walk. the score maximum being 18 (excellent) and minimum 6 (poor)
Rate of Anatomical, Congruent or Incongruent Radiological Outcomes using Matta & Tornetta radiological principles | 1 year postoperative
  Radiological assesment was done according to the grading of Matta and Tornetta, The investigators classified the results into: Anatomical, congruent & incongruent; based on the restoration of the five anatomical lines (iliopectineal line, ilioischial line, acetabular dome, posterior wall & anterior wall) & best judged on the anteroposterior view.
Amount of residual displacement | immediate post-operative and throughout study completion
  Residual displacement was measured in millimeters and compared between the two study groups

SECONDARY OUTCOMES:
post-operative complications' rate | 1-year post-operative
  The investigators focused the evaluation of Postoperative complications on the local complications related to fixation principles and technique: LLD, AVN of the hip joint, wound infection, residual malunion or non-union of the quadrilateral plate, and loss of reduction
Mean intraoperative blood loss | up to 4 days post-operative
  The mean blood loss was calculated and compared between the two study groups, it was measured intraoperative and postoperative from suction drains
Mean operative time | it was calculated intra-operative
  The mean operation time was calculated in minutes and compared between the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Islam S Moussa, MD, Study Chair — no funding recieved
Locations (1):
- Ain Shams university, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
i plan to share it with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one year
Access Criteria: full access